CLINICAL TRIAL: NCT03281629
Title: Circuitry-Guided Smoking Cessation in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Xiaoming Du, Assistant Professsor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HP-00077085; UG3DA047685 (NIH)
Record Dates: First submitted 2017-09-01; First posted 2017-09-13 (Actual); Results first posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Smoking Cessation; Nicotine Addiction; Schizophrenia
Keywords: Transcranial magnetic stimulation; schizophrenia; MRI; smoking
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder; Schizophrenia; Smoking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TMS stimulation (Active Comparator): Real active rTMS stimulation.
  Interventions: Device: Active TMS stimulation
- Sham TMS stimulation (Sham Comparator): Sham repetitive TMS stimulation.
  Interventions: Device: Sham TMS stimulation

INTERVENTIONS:
Device: Active TMS stimulation — Multiple trains of active transcranial magnetic stimulation in a day, for multiple days.
  Arms: Active TMS stimulation
Device: Sham TMS stimulation — Multiple trains of sham transcranial magnetic stimulation in a day, for multiple days.
  Arms: Sham TMS stimulation

SUMMARY:
In a double-blinded, randomized, parallel controlled design, patients with schizophrenia spectrum disorder will be exposed to active or sham repetitive transcranial magentic stimulation (TMS) which was guided by functional magnetic resonance image (MRI). Smoking reduction/cessation and brain functional connectivity changes will be assessed at baseline, different stages of rTMS and/or follow-ups.

DETAILED DESCRIPTION:
Neuroimaging studies suggest that high rate of smoking in patients with schizophrenia may be due to an overlap of nicotine addiction related circuitries and schizophrenia related circuitries, such that schizophrenia impact some of the same circuitries that increase risks for severe nicotine addiction in general. Those identified overlapping circuitries have been linked to several key features of nicotine addiction and can be represented by resting state functional connectivities. Transcranial magnetic stimulation (TMS) provides a non-invasive means for altering brain electrical neural activity. TMS has been approved by FDA for treatment of depression. Other applications have not been approved but it has been used in a wide range of clinical research especially in neurology and psychiatry. There are preliminarily significant improvements in treatments of smoking cessation in schizophrenia using TMS with small samples, but those treatments are not robust in larger samples. The high inter-subject variability limits the efficacy of TMS treatment in schizophrenia patients. We aim to develop a TMS method targeting special brain circuits that are both smoking cessation and schizophrenia related. If the corresponding brain circuits were successfully modulated, the treatment efficacy will be significantly improved and schizophrenia patients will benefit from the TMS treatment of smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female between ages 18-60
* Ability to give written informed consent (age 18 or above)
* Smoking in the last one year or more and average cigarette per day ≥ 5 in the past 4 weeks.
* For patient participants, Evaluation to Sign Consent (ESC) above10.

Exclusion Criteria:

* Any history of seizures
* Had smoking cessation treatment, clinical trial, or nicotine replacements within the past four weeks.
* Significant alcohol or other drug use (substance dependence within 6 months or substance abuse within 1 month) other than nicotine or marijuana dependence.
* Any major medical illnesses that may affect normal brain functioning. Examples of these conditions include, but not limited to, stroke, CNS infection or tumor, other significant brain neurological conditions.
* Taking > 400 mg clozapine/day
* Failed TMS screening questionnaire
* Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
* History of head injury with loss of consciousness over 10 minutes; history of brain surgery
* Can not refrain from using alcohol and/or marijuana 24 hours or more & cigarette smoking one hour or more prior to experiments.
* Woman who is pregnant (child-bearing potential but not on contraceptive and missing menstrual period; or by self report; or by positive pregnancy test).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Du, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fourteen enrolled participants were excluded from the study before assignment to groups. Six of them were excluded because they failed inclusion/exclusion criteria; six of them were excluded due to schedule conflict; one was excluded because the participant cannot fit into MRI scanner; one was excluded because the participant changed mind and decided to quit.
Period: Overall Study
Arm/Group | Active TMS Stimulation | Sham TMS Stimulation
Started | 18 | 12
Completed | 16 | 10
Not Completed | 2 | 2
Not completed — The two participants dropped out due to COVID-19 lockdown. | 2 | 0
Not completed — Death | 0 | 1
Not completed — Participant's schedule change and cannot participate in the study | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TMS Stimulation | Sham TMS Stimulation | Total
Number analyzed (Participants) | 18 | 12 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 12 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (11.8) | 41.9 (12.8) | 43.3 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 11 | 9 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 18 | 11 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 9 | 22
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: Cigarette Per Day
Description: Cigarette per day (CPD) is measured to index smoking reduction and cessation. The change of CPD between baseline and end-of-treatment (1-month time point), 3-month follow up (4-month time point) and 6-month follow up (7-month time point) are reported. Negative values of the change of CPD indicate reductions in cigarette consumption.
Time Frame: 7 months
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Active TMS Stimulation | Sham TMS Stimulation
Number analyzed (Participants) | 18 | 12
cigarettes per day
  Baseline versus End-of-Treatment (1 month) | -3.2 (4.9) | -3.0 (5.1)
  Baseline versus 3-month follow up (4 months time point) | -2.71 (3.10) | -2.50 (3.32)
  Baseline versus 6-month follow up (7 months time point) | -2.50 (2.04) | -3.50 (4.95)

2. Secondary Outcome: Functional Magnetic Resonance Imaging (fMRI)
Description: Resting-state functional connectivity (rsFC) obtained from fMRI is used to evaluate the TMS effect on smoking cessation. The strength of rsFC was first defined by correlation coefficient (r). Because the distribution of r values is highly skewed, z scores (normally distributed) were computed via fisher r-to-z transform. The z score central value (i.e., z score of 0) represents no relationship between the two brain regions. A positive (negative) z score indicates a positive (negative) association between the two brain regions. According to our pilot data determined from a separate study, stronger rsFC (i.e., larger positive z score) was related to less smoking severity. The changes of rsFC between baseline and end-of-treatment (1-month time point) and 3-month follow up (4-month time point) are reported. A positive (negative) value of rsFC change suggests the rsFC was enhanced (weakened) by the intervention. No fMRI data were collected at 6-month follow up (7-month time point).
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: z score of functional connectivity
Arm/Group | Active TMS Stimulation | Sham TMS Stimulation
Number analyzed (Participants) | 18 | 12
z score of functional connectivity
  Baseline versus End-of-Treatment (1 month time point) | 0.025 (0.047) | -0.014 (0.047)
  Baseline versus 3-month follow up (4 months time point) | 0.044 (0.045) | -0.034 (0.011)

3. Secondary Outcome: Cotinine
Description: Cotinine level is an objective index of smoking status. Higher level of cotinine indicates more nicotine consumption. The change of cotinine level between baseline and end-of-treatment (1-month time point) is reported. Cotinine data were not collected at 3-month follow up (4-month time point) or 6-month follow up (7-month time point).
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Active TMS Stimulation | Sham TMS Stimulation
Number analyzed (Participants) | 18 | 12
ng/ml | -112 (1114) | 31 (561)

4. Secondary Outcome: End-expired Carbon Monoxide (CO)
Description: End-expired CO measure is an instant measure of smoking status. Higher CO level indicates more nicotine consumption. The change of CO level between baseline and end-of-treatment (1-month time point) is reported. No CO data were collected at 3-month follow up (4-month time point) or 6-month follow up (7-month time point).
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Active TMS Stimulation | Sham TMS Stimulation
Number analyzed (Participants) | 18 | 12
ppm | -0.67 (9.04) | -2.40 (4.50)

5. Secondary Outcome: Normalized Gamma Power of Auditory Static State Response (ASSR) From Electroencephalography (EEG)
Description: EEG is used to evaluate the brain activities that are corresponding to the TMS. Auditory static state response (ASSR) at gamma frequency (i.e., 40 Hz) is obtained from the EEG recording. The gamma power of ASSR was normalized as the ratio between the power at 40 Hz (i.e., gamma power) and the power of its neighboring frequencies (i.e., 39 and 41 Hz). Increased normalized gamma ASSR is usually related to the improvement of psychosis symptoms. The change of ASSR between baseline and end-of-treatment (1-month time point) and 3-month follow up (4-month time point) are reported. No EEG data were collected at 6-month follow up (7-month time point).
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Active TMS Stimulation | Sham TMS Stimulation
Number analyzed (Participants) | 18 | 12
ratio
  Baseline versus End-pf-Treatment (1 month time point) | 24.0 (37.0) | -38.0 (64.0)
  Baseline versus 3-month follow up (4 months time point) | -5.5 (15.5) | 35.1 (32.8)

ADVERSE EVENTS:
Time Frame: From baseline to the time when the participant completes or quits the study (up to 7 months).
Arm/Group | Active TMS Stimulation | Sham TMS Stimulation
All-Cause Mortality (participants affected / at risk) | 0/18 | 1/12
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/12
Other Adverse Events (participants affected / at risk) | 14/18 | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TMS Stimulation (N=18) | Sham TMS Stimulation (N=12)
Facial muscle twitching (Musculoskeletal and connective tissue disorders) | 8 (8) | 0 (0)
Eye blinks (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
headache (Nervous system disorders) | 4 (4) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 4 (4) | 0 (0)
Uncomfortable click sounds (Ear and labyrinth disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT03281629/Prot_SAP_002.pdf
  • Informed Consent Form (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT03281629/ICF_003.pdf